CLINICAL TRIAL: NCT01172366
Title: A Phase I Study to Evaluate the Potential for Interpersonal Transfer of Testosterone Following Single Dose Application of 2% Testosterone Metered Dose (MD) Lotion®
Brief Title: A Study to Evaluate the Potential for Interpersonal Transfer of Testosterone Following Single Dose Application
Status: Completed | Type: Observational
Sponsor: Acrux DDS Pty Ltd (Industry)
Responsible Party: Director, Clinical Development, Acrux DDS Pty Ltd
Other Study IDs: MTE12
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-08

CONDITIONS: Hypogonadism
Keywords: Open label, single dose, pharmacokinetic study
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The hypotheses for this study is that there is no transfer of testosterone from male (donor) subjects to female (recipient) subjects when contact is made 2 hours post application of 2% Testosterone MD-Lotion® if the donor has a covered application area with a T-shirt.

ELIGIBILITY:
Healthy Male Subjects:

Inclusion:

* Healthy male subjects aged ≥ 18 and ≤ 45, who have no history of clinically significant medical disorders and who have passed the required laboratory and physical screening tests.

Exclusion:

* Men with a history of allergy/sensitivity to testosterone or in whom testosterone therapy is contraindicated, or a clinically significant finding on physical exam or skin disorder.

Healthy Female Subjects:

Inclusion:

* Healthy premenopausal women aged ≥ 18 and ≤ 45, who have no history of clinically significant medical disorders and who have passed the required laboratory and physical screening tests.

Exclusion:

* Women with a history of allergy/sensitivity to testosterone or in whom testosterone therapy is contraindicated, or a clinically significant finding on physical exam or skin disorder.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy male and female volunteers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 72 hours total
  Single dose pharmacokinetic parameters (AUC0-24, AUC0-72, Cmin, Cmax, and tmax) are to be reported for total testosterone, free testosterone and DHT.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Soulis, BSc, PhD, Study Director — Acrux DDS Pty Ltd
Locations (1):
- QPharm, Brisbane, Queensland, Australia